CLINICAL TRIAL: NCT00129779
Title: A Randomised Control Trial Assessing the Effects of an Intermediate Care Package in Preventing Hospitalisation of Elderly Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Assessment of the Effects of an Intermediate Care Package in Preventing Hospitalisation of Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: The Health Foundation (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: NHLICX3038
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2008-05

CONDITIONS: COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Behavioral: Intermediate care package

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a term used for the conditions of chronic bronchitis and emphysema, diseases that are very common among the elderly and diseases that account for up to15% of all general medical admissions to National Health Service Hospitals. In a recent report on emergency admissions to acute hospitals in London, the King's Fund concluded that taking better care of elderly patients with COPD could reduce pressures on acute hospitals, and suggested that identification of vulnerable patients with lung disease and "pro-active," rather than "reactive," management might reduce the chances of hospitalisation. In this study, the investigators wish to compare a group of patients with COPD who are managed in the normal way, with another group of patients with COPD who receive all interventions known to be of some benefit to those with this condition. This will include a pulmonary rehabilitation programme, intensive education regarding self care, targeted advice to their general practitioners regarding how best to manage COPD, and regular contact with specialist respiratory nurses who will support the patients in their own homes by a combination of home visits and telephone contact. The value of such a comprehensive intervention will be studied, in terms of both its ability to reduce admissions to the hospital and its impact on quality of life.

DETAILED DESCRIPTION:
One hundred twenty-two patients over the age of 50 with COPD, admitted to Charing Cross Hospital in 2000-2004 with an acute exacerbation of their condition will be recruited and randomised to routine and opportunistic care (n= 61) vs study care package (n=61) for 2 years. The patients randomised to the study package will take part in an initial pulmonary rehabilitation programme of 8 sessions of physical therapy and education (2 sessions a week for 4 weeks). Health related quality of life will be measured in the intervention and routine care groups using validated instruments (SF-36 and Canadian Respiratory Diseases Questionnaire). This will be followed by a baseline home visit and assessment from an experienced specialist respiratory nurse (Grade G), followed by monthly telephone calls and a home visit every 3 months. Each interview and visit will be a structured intervention addressing specific issues related to the management of COPD, with four possible specific outcomes including history taking; measurement of vital signs; discussion of treatment; appropriate vaccination and discussing and reinforcing self-management education. At the end of the 2 year study period the routine care and intervention groups will be compared for the following outcomes: number of admissions to hospital for exacerbations of COPD; number of unplanned visits to a general practitioner (with those initiated by study nurse identified separately); measures of quality of life (SF-36; CRDQ).

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 50 with COPD
* Admitted to Charing Cross Hospital in 2000-2004 with an acute exacerbation of COPD

Exclusion Criteria:

* Significant co-morbidity including severe heart disease and cancer
* Any condition that would preclude participation in the physical therapy component of a pulmonary rehabilitation programme, including musculoskeletal diseases

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122
Dates: Start 2003-12; Study Completion 2006-08

PRIMARY OUTCOMES:
Number of hospital admissions for exacerbations of COPD

SECONDARY OUTCOMES:
Number of unplanned visits to a general practitioner
Measures of quality of life (SF-36; Canadian Respiratory Disease Questionnaire [CRDQ])

CONTACTS AND LOCATIONS:
Overall Officials: Martyn R Partridge, MD FRCP, Principal Investigator — Imperial College London
Locations (1):
- Respiratory Medicine, NHLI at Charing Cross Hospital, London, United Kingdom

REFERENCES:
- [Background] The burden of lung disease. British Thoracic Society, London, 2001.
- [Background] King's Fund report - 'Managing the pressure' by Michael Damiani and Jennifer Dixon. King's Fund, London 2002
- [Background] Gravil JH, Al-Rawas OA, Cotton MM, Flanigan U, Irwin A, Stevenson RD. Home treatment of exacerbations of chronic obstructive pulmonary disease by an acute respiratory assessment service. Lancet. 1998 Jun 20;351(9119):1853-5. doi: 10.1016/s0140-6736(97)11048-0. PMID 9652670
- [Background] Cockcroft A, Bagnall P, Heslop A, Andersson N, Heaton R, Batstone J, Allen J, Spencer P, Guz A. Controlled trial of respiratory health worker visiting patients with chronic respiratory disability. Br Med J (Clin Res Ed). 1987 Jan 24;294(6566):225-8. doi: 10.1136/bmj.294.6566.225. PMID 3101821
- [Background] Lacasse Y, Wong E, Guyatt GH, King D, Cook DJ, Goldstein RS. Meta-analysis of respiratory rehabilitation in chronic obstructive pulmonary disease. Lancet. 1996 Oct 26;348(9035):1115-9. doi: 10.1016/S0140-6736(96)04201-8. PMID 8888163
- [Background] British Thoracic Society Standards of Care Subcommittee on Pulmonary Rehabilitation. Pulmonary rehabilitation. Thorax. 2001 Nov;56(11):827-34. doi: 10.1136/thorax.56.11.827. No abstract available. PMID 11641505
- [Background] Parrott S, Godfrey C, Raw M, West R, McNeill A. Guidance for commissioners on the cost effectiveness of smoking cessation interventions. Thorax. 1998 Dec;53 Suppl 5 Pt 2(Suppl 5):S1-38. No abstract available. PMID 10226676
- [Background] Raw M, McNeill A, Watt J, Raw D. National smoking cessation services at risk. BMJ. 2001 Nov 17;323(7322):1140-1. doi: 10.1136/bmj.323.7322.1140. No abstract available. PMID 11711385
- [Background] Gallefoss F, Bakke PS. Impact of patient education and self-management on morbidity in asthmatics and patients with chronic obstructive pulmonary disease. Respir Med. 2000 Mar;94(3):279-87. doi: 10.1053/rmed.1999.0749. PMID 10783940
- [Background] BTS guidelines for the management of chronic obstructive pulmonary disease. The COPD Guidelines Group of the Standards of Care Committee of the BTS. Thorax. 1997 Dec;52 Suppl 5(Suppl 5):S1-28. No abstract available. PMID 9474238
- [Background] Pauwels RA, Buist AS, Calverley PM, Jenkins CR, Hurd SS; GOLD Scientific Committee. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease. NHLBI/WHO Global Initiative for Chronic Obstructive Lung Disease (GOLD) Workshop summary. Am J Respir Crit Care Med. 2001 Apr;163(5):1256-76. doi: 10.1164/ajrccm.163.5.2101039. No abstract available. PMID 11316667
- [Derived] Sridhar M, Taylor R, Dawson S, Roberts NJ, Partridge MR. A nurse led intermediate care package in patients who have been hospitalised with an acute exacerbation of chronic obstructive pulmonary disease. Thorax. 2008 Mar;63(3):194-200. doi: 10.1136/thx.2007.077578. Epub 2007 Sep 27. PMID 17901162